CLINICAL TRIAL: NCT02668523
Title: A Prospective, Multicenter Clinical Trial to Evaluate the Safety and Effectiveness of the ReVision Optics, Inc., RAINDROP® NEAR VISION INLAY for the Improvement of Near and Intermediate Vision in Pseudophakic Subjects
Brief Title: A Clinical Trial to Evaluate a Corneal Inlay for the Improvement of Near and Intermediate Vision in Pseudophakic Presbyopic Subjects
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ReVision Optics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P15-0010
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Presbyopia; Pseudophakia
Keywords: Presbyopia; Corneal Inlay; Pseudophakic; Pseudophakia
MeSH Terms: conditions — Presbyopia; Pseudophakia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Raindrop (Experimental): A single arm study to evaluate the effectiveness of a 2mm Raindrop Near Vision Inlay for the treatment of presbyopia in pseudophakic subjects. This corneal inlay is placed under a LASIK flap or in a corneal pocket, and is designed to change the anterior curvature of the cornea, resulting in the ability to reduce spectacle dependency for near and intermediate tasks.
  Interventions: Device: Raindrop Near Vision Inlay

INTERVENTIONS:
Device: Raindrop Near Vision Inlay — To improve the near and intermediate vision in subjects who have previously undergone cataract surgery (pseudophakic subjects)

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the Raindrop Near Vision Inlay implanted in bilateral pseudophakes with presbyopia for improvement of near and intermediate vision.

DETAILED DESCRIPTION:
The loss of near vision and the ability to perform tasks that require near vision is part of the normal aging process. This natural transformation in the eye occurs as a result of the loss of accommodation of the crystalline lens, a condition known as presbyopia. Presbyopia, characterized by a progressive, age-related loss of accommodation (i.e., the lens ability to focus clearly over a wide range of distances), is most prevalent of all visual deficiencies, affecting 100% of the population over the course of a normal life span.

Presbyopia is also a natural outcome of pseudophakic subjects with monofocal or toric intraocular lenses. Treatment of pseudophakic presbyopia generally consists of reading glasses, contact lenses, or monovision LASIK which allows the patient to see near objects. All these options present limitations from the patient perspective.

ReVision Optics has developed the Raindrop corneal inlay for the correction of near vision. The Raindrop is a 2mm corneal inlay, as small as a pinhead, thinner than a human hair and about 1/500th of a droplet of water. The inlay is the same refractive index as the human cornea. The inlay is placed in the non-dominant eye, centered over the pupil after a corneal flap or corneal pocket has been made. The Raindrop is expected to provide pseudophakic presbyopic subjects with improvement of near and intermediate vision.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide informed consent, have signed the written informed consent form, and been given a copy.
2. Subjects must be bilateral pseudophakic adults with presbyopia, needing reading add from +1.50 D to +2.50 D.
3. Subjects must be at least 50 years old
4. Subjects must have uncorrected near visual acuity worse than 20/40 and better than 20/200 in the non-dominant eye.
5. Subjects must have monocular uncorrected distance visual acuity of 20/25 or better in both eyes.
6. Subjects must have distance and near visual acuity correctable to at least 20/20 in both eyes.
7. Subjects must have a manifest refraction spherical equivalent (MRSE) between -0.50 and +1.00 D with no more than 0.75 D of refractive cylinder in the non-dominant eye.
8. Subjects must have a tear break-up time (TBUT) of ≥8 seconds.
9. Subjects must have a central corneal thickness of between 480 and 600 microns in the non-dominant eye.
10. Subjects must have an average corneal power of ≥ 41.00 D and ≤ 47.00 D in the non-dominant eye.
11. Subjects must have a photopic pupil size of ≥3.0 mm, in the non-dominant eye.
12. Subjects must have an endothelial cell count ≥ 2200 cells/mm2 in the eye to be implanted (non-dominant).
13. Subjects who are contact lens wearers must discontinue hard or rigid gas permeable lenses for at least 3 weeks and discontinue soft lenses for at least 1 week prior to baseline examination.
14. Subjects who are contact lens wearers must have two (2) central keratometry readings with regular mires and two (2) manifest refractions taken at least one week apart, with no contact lens wear between. Keratometric values must not differ by more than ± 0.50 D in any meridian the eye to be implanted. MRSE values must not differ more than ±0.50 D in the non-dominant eye.
15. Subjects must have documented monovision tolerance as determined by a 5-day contact lens trial prior to surgery.
16. Subjects must have a minimum of 3 months between cataract surgery and implantation of the Raindrop Near Vision Inlay in the non-dominant eye.
17. Subjects must be able to demonstrate refractive stability after cataract surgery (e.g., No change in MRSE greater than ± 0.50 D within the last 2 consecutive visual examinations after IOL implantation, performed at least 3 months apart.
18. Subjects must have a clear or open posterior capsule in the non-dominant eye.
19. Subjects must be willing and able to return for scheduled follow-up examinations for 24 months after surgery.

Exclusion Criteria:

1. Subjects with anterior chamber or multifocal IOLs (intraocular lens) in either eye.
2. Subjects with clinically significant anterior segment pathology in either eye.
3. Subjects who have worn soft or rigid contact lenses within the past 30 days in the eye to be treated (excludes the contact lens trial for monovision tolerance).
4. Subjects with residual, recurrent, active ocular or uncontrolled eyelid disease (e.g., meibomian gland dysfunction), or any corneal abnormality (including endothelial dystrophy, guttata, recurrent corneal erosion, etc.) in either eye.
5. Subjects with ophthalmoscopic signs of keratoconus (or keratoconus suspect) in either eye.
6. Subjects with distorted or unclear corneal mires on topography maps of the non- dominant eye.
7. Subjects who require canthotomy to generate a corneal flap in the non-dominant eye.
8. Subjects with macular degeneration, retinal detachment, or any other fundus pathology that would prevent an acceptable visual outcome in either eye.
9. Subjects who have undergone previous corneal surgery including LASIK surgery in the non-dominant eye.
10. Subjects with a history of ocular herpes zoster or ocular herpes simplex keratitis.
11. Subjects who have a history of steroid-responsive rise in intraocular pressure, preoperative IOP > 21 mm Hg, glaucoma, or who are a glaucoma suspect in either eye.
12. Subjects with a history of uncontrolled diabetes, autoimmune disease, connective tissue disease, or clinically significant atopic syndrome.
13. Subjects on chronic systemic corticosteroids or other immunosuppressive therapy that may affect wound healing, and any immunocompromised subjects.
14. Subjects who are using ophthalmic medication(s) other than artificial tears for treatment of any ocular pathology excluding ocular allergy.
15. Subjects using systemic medications with significant ocular side effects.
16. Subjects with known sensitivity to planned study concomitant medications.
17. Subjects who are participating in any other clinical trial during the course of this clinical investigation.
18. Subjects who have had previous astigmatic keratotomy or limbal relaxing incisions at the time of cataract surgery.
19. Subjects who are of child bearing potential and who have a positive pregnancy test result, prior to surgery.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-03 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Improvement in uncorrected near visual acuity | 24 Months
  Seventy-five percent of eyes should achieve uncorrected near visual acuity of 20/40 or better.
Preservation of best corrected visual acuity | 24 Months
  Fewer than five percent of eyes should lose more than 2 lines of best corrected distance visual acuity after implantation

SECONDARY OUTCOMES:
Improvement in uncorrected intermediate visual acuity | 24 Months
  Seventy-five percent of eyes should achieve uncorrected intermediate visual acuity of 20/40 or better (measured at 80cm/32 inches)
Adverse Events | 24 Months
  Adverse events should occur in less than 10% of eyes and any single adverse event should occur in less than 2.5% of eyes.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Harvard Eye Associates, Laguna Hills, California
  - Coastal Vision Laser Eye Center, Orange, California
  - The Eye Associates of Manatee, Bradenton, Florida
  - The Eye Institute of West Florida, Largo, Florida
  - The Bowie Vision Institute, Bowie, Maryland
  - Chu Vision Institute, Bloomington, Minnesota
  - Associated Eye Care, Stillwater, Minnesota
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Key-Whitman Eye Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Parkhurst NuVision, San Antonio, Texas
  - The Eye Institute of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No